CLINICAL TRIAL: NCT01521507
Title: Randomized Controlled Trial of Long-term Treatment Effectiveness for Meibomian Gland Dysfunction (MGD) and Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TearScience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LF-004
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Meibomian Gland Dysfunction; Dry Eye
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LipiFlow System (Experimental): Treatment with LipiFlow System at randomization in Stage 1 of study
  Interventions: Device: LipiFlow System
- Warm Compress and Lid Hygiene (Active Comparator): Control group receiving warm compress therapy and lid hygiene at randomization in Stage 1 of study and crossover LipiFlow System treatment in Stage 2 of study
  Interventions: Device: LipiFlow System; Device: Warm Compress Therapy + Lid Scrub

INTERVENTIONS:
Device: LipiFlow System — In-office device treatment for meibomian gland dysfunction by a physician
Device: Warm Compress Therapy + Lid Scrub — At-home daily warm compress therapy and lid hygiene
  Other Names: EyeGiene Warm Compress Therapy; OCuSOFT Lid Scrub
  Arms: Warm Compress and Lid Hygiene

SUMMARY:
The study objective is to evaluate the long-term treatment effectiveness for adult patients with meibomian gland dysfunction (MGD) and evaporative dry eye by: 1) comparing the LipiFlow® System to a standardized daily warm compress and eyelid hygiene control therapy over a duration of 3 Months; and 2) evaluating the LipiFlow® alone and in combination with other MGD and dry eye treatments over a duration of up to 12 Months.

This is a post-market, non-significant risk, prospective and multi-center clinical trial divided into two stages. The first stage from enrollment to 3 Months is an open-label, randomized controlled design to compare the effectiveness of a single LipiFlow® System treatment to a standardized daily warm compress and eyelid hygiene Control therapy with Crossover LipiFlow® treatment of the Control subjects at 3 Months. The second stage, occurring between 3 and 12 Months, is an observational design to evaluate the effectiveness of LipiFlow® alone and in combination with other MGD and dry eye treatments over a duration of up to 12 Months. Subjects are entered into the following subgroups based on the subject's self-assessment of the adequacy of symptom relief and protocol-defined criteria for additional treatment.

1. One LipiFlow® Treatment: Subjects who receive only one LipiFlow® treatment.
2. Two LipiFlow® Treatments: Subjects who receive a second LipiFlow® treatment.
3. Combination Treatment: Subjects who receive one or two LipiFlow® treatments followed by other MGD or dry eye treatment, as prescribed by the physician.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Tear film assessment that qualifies in both eyes
* Evidence of meibomian gland dysfunction and dry eye in both eyes
* Willingness to comply with study protocol

Exclusion Criteria:

* Systemic disease condition or medication that causes dry eye
* Use of other treatments for MGD or dry eye
* Ocular surgery, trauma, herpes infection, punctal plug insertion or punctal occlusion within past 3 months
* Active eye infection
* Active eye inflammation or recurrent inflammation within past 3 months
* Moderate to severe allergic conjunctivitis
* Severe eyelid inflammation
* Eyelid abnormality that affects lid function
* Ocular surface abnormality that may compromise corneal integrity
* Pregnant or nursing women
* Participation in another ophthalmic clinical trial within past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-01; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christy Stevens, O.D., Study Director — TearScience, Inc.
Locations (9):
- United States (9):
  - McDonald Eye Associates, Fayetteville, Arkansas
  - Harvard Eye Associates, Laguna Hills, California
  - Center for Excellence in Eye Care, Miami, Florida
  - Chicago Cornea Consultants, Ltd., Hoffman Estates, Illinois
  - Jackson Eye, Lake Villa, Illinois
  - Cincinnati Eye Institute - Northern Kentucky, Edgewood, Kentucky
  - Charles River Eye Associates, Winchester, Massachusetts
  - Associated Eye Care, Stillwater, Minnesota
  - Ophthalmology Consultants, Ltd., St Louis, Missouri

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 19, 2012 and October 15, 2012, this study enrolled subjects with meibomian gland dysfunction (MGD) and evaporative dry eye from nine ophthalmic practices in the United States.
Pre-assignment Details: A total of 274 subjects were consented and 200 subjects were randomized. Of the 74 subjects who were not randomized, 52 subjects did not meet the study eligibility criteria and 22 subjects elected not to participate prior to randomization or had not yet attended the Baseline visit when study enrollment was completed.
Groups:
- LipiFlow Treatment: Subjects received a single, 12-minute, in-office treatment of both eyes for MGD with the LipiFlow System after randomization in Stage 1 of study.
  In Stage 2, subjects were entered into subgroups based on the subject's assessment of adequacy of symptom relief:
  1. One LipiFlow Treatment - After subjects received one LipiFlow treatment at randomization, no other MGD or dry eye treatment was prescribed for the study duration.
  2. Two LipiFlow Treatments - Subjects received a second LipiFlow treatment during Stage 2. No other MGD or dry eye treatment was prescribed for the study duration.
  3. Combination Treatment - After subjects received one or two LipiFlow treatments, they received other MGD or dry eye treatment, as prescribed by the physician.
- Warm Compress & Lid Hygiene, Then Crossover LipiFlow Treatment: Subjects received twice-daily, standardized warm compress therapy and lid hygiene in both eyes from randomization to 3 months in Stage 1. Then, subjects received a single, 12-minute crossover LipiFlow treatment of both eyes.
  In Stage 2, subjects were entered into subgroups based on the subject's assessment of adequacy of symptom relief:
  1. One LipiFlow Treatment - After subjects received one LipiFlow treatment at crossover, no other MGD or dry eye treatment was prescribed for the study duration.
  2. Two LipiFlow Treatments - Subjects received a second LipiFlow treatment during Stage 2. No other MGD or dry eye treatment was prescribed for the study duration.
  3. Combination Treatment - After subjects received one or two LipiFlow treatments, they received other MGD or dry eye treatment, as prescribed by the physician.
Period: Stage 1: Randomized Design
Arm/Group | LipiFlow Treatment | Warm Compress & Lid Hygiene, Then Crossover LipiFlow Treatment
Started | 101 | 99
Received Initial Treatment (Tx) | 99 | 98
Completed | 98 | 94
Not Completed | 3 | 5
Not completed — Device did not fit, No Treatment | 2 | 0
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 0 | 2
Period: Stage 2: Observational Design
Arm/Group | LipiFlow Treatment | Warm Compress & Lid Hygiene, Then Crossover LipiFlow Treatment
Started | 98 | 94
Received Crossover LipiFlow Tx | 0 | 93
Received Only One LipiFlow Tx at 12 Mo | 81 | 82
Received Other MGD Treatment at 12 Mo | 11 | 9
Received 2nd LipiFlow Tx at 12 Mo | 2 | 1
Completed | 94 | 92
Not Completed | 4 | 2
Not completed — Device did not fit, No Treatment | 0 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- LipiFlow Treatment: Subjects received a single, 12-minute, in-office treatment of both eyes for MGD with the LipiFlow System after randomization in Stage 1 of study.
- Warm Compress & Lid Hygiene: Subjects received twice-daily, standardized warm compress therapy and lid hygiene in both eyes from randomization to 3-month visit in Stage 1.
- Total: Total of all reporting groups
Arm/Group | LipiFlow Treatment | Warm Compress & Lid Hygiene | Total
Number analyzed (Participants) | 101 | 99 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (15.9) | 56.1 (14.7) | 56.2 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 68 | 142
  Male | 27 | 31 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 14
  Not Hispanic or Latino | 94 | 92 | 186
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 98 | 96 | 194
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 101 | 99 | 200
Baseline Total Meibomian Gland Score [Mean (Standard Deviation); unit: units on a scale] | 6.2 (3.7) | 6.3 (3.7) | 6.2 (3.7)
Baseline Total OSDI Score [Mean (Standard Deviation); unit: units on a scale] | 45.6 (21.2) | 51.8 (23.1) | 48.7 (22.4)
Duration of Dry Eye Symptoms [Mean (Standard Deviation); unit: years] | 6.9 (6.8) | 8.7 (7.7) | 7.8 (7.3)
Duration of MGD or Dry Eye Diagnosis [Mean (Standard Deviation); unit: years] | 5.3 (6.2) | 5.5 (5.9) | 5.4 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Stage 1 Mean Change in Total Meibomian Gland Score From Baseline to 3 Months
Description: To assess the meibomian glands, the secretion characteristics from 15 gland orifices along the lower eyelid were evaluated under a slit lamp biomicrosope using a handheld instrument, Meibomian Gland Evaluator, to apply gentle standardized pressure to the eyelid margin. Expressed secretion characteristics were graded on a scale of 3 (clear liquid secretion), 2 (cloudy liquid secretion), 1 (inspissated/toothpaste consistency), and 0 (no secretion). Total meibomian gland score was calculated based on the sum of the secretion grades for all 15 glands over a range from 0 to 45 with a higher score reflecting less meibomian gland dysfunction. To be eligible for the study, the Baseline total meibomian gland score must have been 12 or less in each eye. Change = 3 Month score - Baseline Score.
Time Frame: Baseline and 3 Months
Population: Intent to Treat Population (All Participants who were randomized and received at least partial LipiFlow treatment or used warm compress therapy at least once and had data available at 3 Months).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | LipiFlow Treatment | Warm Compress & Lid Hygiene
Number analyzed (Participants) | 98 | 94
units on a scale | 11.6 [10.2 to 13.0] | 4.5 [3.4 to 5.6]
Statistical Analysis 1: Comparison: LipiFlow Treatment vs Warm Compress & Lid Hygiene; The null and alternative hypotheses are H0: µt ≤ µc vs. Ha: µt > µc, where µt and µc are the mean changes in total meibomian gland scores from Baseline to 3 Months for the LipiFlow (test) and Warm Compress and Lid Hygiene (active control) groups, respectively. For the Stage 1 Primary Outcome, the minimum sample size was 24 subjects per group with a power of 90% and a one-sided alpha of 0.025; Test type: Superiority or Other; p < 0.0001, z-statistic — Stage 1 primary and secondary outcomes were tested in order under a closed form testing method. Secondary outcome was tested only if primary outcome was statistically significant. If both outcomes were significant, overall study alpha was 0.025; p-value was based on z-statistic of the sum of weighted average of difference in scores between groups at each site divided by the sum of the weights
Statistical Analysis 2: Comparison: LipiFlow Treatment vs Warm Compress & Lid Hygiene; Supportive multivariate mixed model was also performed for this outcome controlling for significant demographic and baseline characteristics; Test type: Superiority or Other; p = 0.0020, Mixed Models Analysis

2. Primary Outcome: Stage 2 Mean Total Meibomian Gland Score at 12 Months
Description: To assess the meibomian glands, the secretion characteristics from 15 gland orifices along the lower eyelid were evaluated under a slit lamp biomicrosope using a handheld instrument, Meibomian Gland Evaluator, to apply gentle standardized pressure to the eyelid margin. Expressed secretion characteristics were graded on a scale of 3 (clear liquid secretion), 2 (cloudy liquid secretion), 1 (inspissated/toothpaste consistency), and 0 (no secretion). Total meibomian gland score was calculated based on the sum of the secretion grades for all 15 glands over a range from 0 to 45 with a higher score reflecting less meibomian gland dysfunction. The total meibomian gland score at 12 Months was compared across subgroups, as defined below.
Time Frame: 12 Months
Population: Intent to Treat Population (All participants who received at least partial LipiFlow or Crossover LipiFlow treatment and had data available at 12 Months). Two LipiFlow treatments subgroup was not analyzed because sample size was too small (n<5) for meaningful analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- LipiFlow Arm: One LipiFlow Treatment Subgroup: Subjects received a single, 12-minute, in-office LipiFlow treatment of both eyes after randomization in Stage 1.
  In Stage 2, subjects were entered into subgroups based on the subject's assessment of adequacy of symptom relief. In the One LipiFlow Treatment subgroup, no other MGD or dry eye treatment was prescribed for the study duration.
- LipiFlow Arm: Combination Treatment Subgroup: Subjects received a single, 12-minute, in-office LipiFlow treatment of both eyes after randomization in Stage 1.
  In Stage 2, subjects were entered into subgroups based on the subject's assessment of adequacy of symptom relief. In the Combination Treatment subgroup, subjects received one LipiFlow treatment (at randomization) followed by other MGD or dry eye treatment, as prescribed by the physician.
- Warm Compress/Hygiene Arm: One LipiFlow Treatment Subgroup: After 3 months of using standardized warm compress therapy and lid hygiene, subjects received a single, 12-minute crossover LipiFlow treatment of both eyes.
  In Stage 2, subjects were entered into subgroups based on the subject's assessment of adequacy of symptom relief. In the One LipiFlow Treatment subgroup, no other MGD or dry eye treatment was prescribed for the study duration.
- Warm Compress/Hygiene Arm: Combination Treatment Subgroup: After 3 months of using standardized warm compress therapy and lid hygiene, subjects received a single, 12-minute crossover LipiFlow treatment of both eyes.
  In Stage 2, subjects were entered into subgroups based on the subject's assessment of adequacy of symptom relief. In the Combination Treatment subgroup, subjects received one LipiFlow treatment (at crossover) or two LipiFlow treatments followed by other MGD or dry eye treatment, as prescribed by the physician.
Arm/Group | LipiFlow Arm: One LipiFlow Treatment Subgroup | LipiFlow Arm: Combination Treatment Subgroup | Warm Compress/Hygiene Arm: One LipiFlow Treatment Subgroup | Warm Compress/Hygiene Arm: Combination Treatment Subgroup
Number analyzed (Participants) | 81 | 11 | 82 | 9
units on a scale | 17.3 [15.8 to 18.7] | 17.9 [13.1 to 22.7] | 18.4 [16.7 to 20.1] | 17.4 [13.2 to 21.6]
Statistical Analysis 1: Comparison: LipiFlow Arm: One LipiFlow Treatment Subgroup vs LipiFlow Arm: Combination Treatment Subgroup vs Warm Compress/Hygiene Arm: One LipiFlow Treatment Subgroup vs Warm Compress/Hygiene Arm: Combination Treatment Subgroup; The null and alternative hypotheses for the Stage 2 Primary Outcome was: H0: µi= µj for all i and j where i≠j versus Ha: µi ≠ µj for at least one i and j, where µi is the mean total meibomian gland score at 12 Months for the ith subgroup. The null hypothesis was tested with a two-sided test at alpha=0.05. Since Stage 2 was an observational design, no minimum sample size was calculated for Stage 2; Test type: Superiority or Other; p = 0.9098, Mixed Models Analysis; Stage 2 Primary Outcome was analyzed with a multivariate mixed model with the subgroup as a fixed effect while controlling for other covariates

3. Secondary Outcome: Stage 1 Mean Change in Total OSDI Score From Baseline to 3 Months
Description: Dry eye symptoms assessed using the OSDI questionnaire were sensitivity to light, grittiness, pain or soreness, blurred vision and poor vision. The questionnaire evaluated the frequency problems with the eyes limited performance in reading, driving at night, working with a computer or bank machine, and watching television. Also, the frequency that eyes felt uncomfortable was assessed in windy conditions, areas with low humidity, and air-conditioned areas. The frequency scale was 0 (none of the time), 1 (some of the time), 2 (half of the time), 3 (most of the time), and 4 (all of the time). The total OSDI score was calculated as the sum of frequency scores for all symptoms multiplied by 25 and divided by the number of questions answered with a range from 0 to 100. A lower total OSDI score represents less disability from dry eye symptoms. To be eligible for the study, the Baseline total OSDI score must have been 13 points or higher in each eye. Change=3 Months score-Baseline score.
Time Frame: Baseline, 3 Months
Population: Intent to Treat Population (All participants who were randomized and received at least partial device treatment or used warm compress at least once and had data available at 3 Months).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | LipiFlow Treatment | Warm Compress & Lid Hygiene
Number analyzed (Participants) | 98 | 94
units on a scale | -23.4 [-26.3 to -20.5] | -17.8 [-20.7 to -14.9]
Statistical Analysis 1: Comparison: LipiFlow Treatment vs Warm Compress & Lid Hygiene; The null and alternative hypotheses are H0: µt ≤ µc vs. Ha: µt > µc, where µt and µc are the mean changes in total OSDI scores from Baseline to 3 Months for the LipiFlow (test) and Warm Compress and Lid Hygiene (active control) groups, respectively. For the Stage 1 Secondary Outcome, the minimum sample size was 84 per group with a power of 80% and a one-sided alpha of 0.025; Test type: Superiority or Other; p = 0.0068, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: LipiFlow Treatment vs Warm Compress & Lid Hygiene; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0419, Mixed Models Analysis

4. Secondary Outcome: Stage 2 Mean Total OSDI Score at 12 Months
Description: Dry eye symptoms assessed using the OSDI questionnaire were sensitivity to light, grittiness, pain or soreness, blurred vision and poor vision. The questionnaire evaluated the frequency problems with the eyes limited performance in reading, driving at night, working with a computer or bank machine, and watching television. Also, the frequency that eyes felt uncomfortable was assessed in windy conditions, areas with low humidity, and air-conditioned areas. Frequency scale was 0 (none of the time), 1 (some of the time), 2 (half of the time), 3 (most of the time), and 4 (all of the time). The total OSDI score was calculated as the sum of frequency scores for all symptoms multiplied by 25 and divided by the number of questions answered with a range from 0 to 100. A lower total OSDI score represents less disability from dry eye symptoms. The total OSDI score at 12 Months was compared across subgroups, as defined below.
Time Frame: 12 Months
Population: Intent to Treat (All participants who received at least a partial LipiFlow treatment or Crossover LipiFlow treatment and had data available at 12 Months). The Two LipiFlow treatments subgroup was not analyzed because the sample size (n<5) was too small for meaningful analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- LipiFlow Arm: One LipiFlow Treatment Subgroup: Subjects received a single, 12-minute, in-office treatment of both eyes for MGD with the LipiFlow System after randomization in Stage 1 of study.
  In Stage 2, subjects were entered into subgroups based on the subject's assessment of adequacy of symptom relief. In the One LipiFlow Treatment subgroup, no other MGD or dry eye treatment was prescribed for the study duration.
- LipiFlow Arm: Combination Treatment Subgroup: Subjects received a single, 12-minute, in-office treatment of both eyes for MGD with the LipiFlow System after randomization in Stage 1 of study.
  In Stage 2, subjects were entered into subgroups based on the subject's assessment of adequacy of symptom relief. In the Combination Treatment subgroup, subjects received one LipiFlow treatment (at randomization) followed by other MGD or dry eye treatment, as prescribed by the physician.
Arm/Group | LipiFlow Arm: One LipiFlow Treatment Subgroup | LipiFlow Arm: Combination Treatment Subgroup | Warm Compress/Hygiene Arm: One LipiFlow Treatment Subgroup | Warm Compress/Hygiene Arm: Combination Treatment Subgroup
Number analyzed (Participants) | 81 | 11 | 82 | 9
units on a scale | 21.6 [18.3 to 24.9] | 35.8 [24.5 to 47.1] | 24.0 [20.5 to 27.6] | 42.2 [25.5 to 58.9]
Statistical Analysis 1: Comparison: LipiFlow Arm: One LipiFlow Treatment Subgroup vs LipiFlow Arm: Combination Treatment Subgroup vs Warm Compress/Hygiene Arm: One LipiFlow Treatment Subgroup vs Warm Compress/Hygiene Arm: Combination Treatment Subgroup; The null and alternative hypotheses for the Stage 2 Secondary Outcome was: H0: µi= µj for all i and j where i≠j versus Ha: µi ≠ µj for at least one i and j, where µi is the mean total OSDI score at 12 Months for the ith subgroup. The null hypothesis was tested with a two-sided test at alpha=0.05. Since Stage 2 was an observational design, no minimum sample size was calculated for Stage 2; Test type: Superiority or Other; p = 0.0237, Mixed Models Analysis — Stage 2 Secondary Outcome was analyzed with a multivariate mixed model with the subgroup as a fixed effect while controlling for other covariates

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 1 year.
Description: Device-related adverse events were evaluated by arm/group. Events occurring during Stage 1 were assessed based on relationship to the LipiFlow Treatment or Warm Compress Therapy and Lid Hygiene. Events occurring in Stage 2 were assessed based on relationship to LipiFlow Treatment or Crossover LipiFlow Treatment.
Groups:
- Crossover LipiFlow Treatment: After using twice-daily, standardized warm compress therapy and lid hygiene for 3 months, subjects received a single, 12-minute crossover LipiFlow treatment of both eyes.
Arm/Group | LipiFlow Treatment | Warm Compress & Lid Hygiene | Crossover LipiFlow Treatment
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/99 | 0/94
Other Adverse Events (participants affected / at risk) | 6/101 | 7/99 | 4/94
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LipiFlow Treatment (N=101) | Warm Compress & Lid Hygiene (N=99) | Crossover LipiFlow Treatment (N=94)
Anterior Staphylococcal Blepharitis (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Blurry Vision (Eye disorders) | 1 (1) | 1 (2) | 0 (0)
Burning Sensation (Eye disorders) | 0 (0) | 1 (2) | 1 (2)
Chalazion (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye/Eyelid Discomfort/Pain (Eye disorders) | 3 (4) | 1 (2) | 1 (2)
Eyelid Edema/Swelling (Eye disorders) | 1 (2) | 1 (2) | 1 (2)
Eyelid Erythema/Redness (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Eyelid Irritation (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Eyelid Itching (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Eyelid Dermatitis (Eye disorders) | 0 (0) | 2 (3) | 0 (0)
Flashes/Ocular Migraine (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Gritty Sensation (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Hordeolum (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Increase/Worsening of MGD (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Increase/Worsening of Ocular Dryness (Eye disorders) | 0 (0) | 1 (2) | 2 (4)
Photophobia/Light Sensitivity (Eye disorders) | 0 (0) | 1 (2) | 1 (1)
Tearing (Eye disorders) | 0 | 1 (2) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review communications for at least 30 days prior to public release with an extension for up to 45 additional days, if the Sponsor notifies the Investigator that the publication contains patentable material or Proprietary Information other than the study results. Upon Sponsor's written request, Investigator agrees to delete any Proprietary Information.